CLINICAL TRIAL: NCT05215639
Title: Venetoclax AML Observational Real-World Study of Treatment-naïve Patients Ineligible for Intensive Chemotherapy in Switzerland & Austria
Brief Title: A Study to Assess Change in Disease State in Adult Participants With Acute Myeloid Leukemia (AML) Ineligible for Intensive Chemotherapy in Switzerland and Austria Receiving Oral Venetoclax Tablets
Acronym: VALOR
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P21-937
Record Dates: First submitted 2022-01-19; First posted 2022-01-31 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Venetoclax; Venclexta; Venclyxto; ABT-199; Cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Venetoclax Participants: Participants treated with Venetoclax in accordance with approved local label.

SUMMARY:
Acute myeloid leukemia (AML) is a cancer of the blood and bone marrow and is the most common acute leukemia in adults. This study will evaluate how well Venetoclax works to treat AML in adult participants who are ineligible for intensive chemotherapy in Switzerland & Austria.

Venetoclax is a drug approved to treat acute myeloid leukemia. All study participants will receive Venetoclax as prescribed by their study doctor in accordance with approved local label. Adult participants with a new diagnosis of AML who are ineligible for intensive chemotherapy will be enrolled. Around 120 participants will be enrolled in the study in approximately 15 sites in Switzerland & Austria.

Participants will receive venetoclax tablets to be taken by mouth daily according to the approved local label. The duration of the study is approximately 24 months.

There is expected to be no additional burden for participants in this trial. All study visits will occur during routine clinical practice and participants will be followed for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed AML and eligible to receive venetoclax as per local label.
* Physician has decided to initiate venetoclax treatment. The decision to treat with venetoclax is made by the physician in accordance with the local label prior to any decision to approach the patient to participate in this study.

Exclusion Criteria:

- Participating in an interventional clinical trial within 30 days prior to venetoclax treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with acute myeloid leukemia (AML) treated with Venetoclax per approved local label in Switzerland & Austria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Overall Survival (OS) | Up to Month 24
  OS is defined as the time from treatment initiation to death from any cause.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Composite Complete Remission | Up to Month 24
  Composite complete remission is defined as the proportion of participants with complete remission (CR) or complete remission with incomplete marrow recovery (CRi).
Time to Transfusion Independence | Up to Month 24
  Time to transfusion independence is defined as the time between the date of first venetoclax intake and the absence of any Red Blood Cell (RBC) or platelet transfusion during any consecutive 8 and/or 16 weeks during the treatment period and percentage of participants achieving transfusion independence.
Change from Baseline in European Quality of Life 5 Dimensions (EQ-5D-5L) Considered Minimally Clinical Important | Up to Month 24
  The EQ-5D-5L is a standardized instrument used to measure health-related quality of life that can be used in a wide range of health conditions and treatments.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Considered Minimally Clinical Important | Up to Month 24
  The EORTC QLQ-C30 is developed to assess the quality of life of cancer patients and is based on multi-item and single-item scales. The core questionnaire contains 5 functional scales, 3 symptom scales, 1 global health status scale, as well as 6 single-item measures.
Treatment Patterns Venetoclax in Combination with Hypomethylating Agents (HMAs) and in Switzerland in combination with Low Dose Cytarabine (LDAC) | Up to Month 24
  Treatment patterns defined by the proportion of participants treated with venetoclax in combination with HMAs and in Switzerland in combination with LDAC.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (19):
- Austria (7):
  - Klinikum Klagenfurt am Wörthersee /ID# 247304, Klagenfurt, Carinthia
  - Universitaetsklinikum St. Poelten /ID# 247283, Sankt Pölten, Lower Austria
  - Krankenhaus der Barmherzigen Brueder Graz /ID# 254121, Graz, Styria
  - Landeskrankenhaus Hochsteiermark, Standort Leoben /ID# 254174, Leoben, Styria
  - Ordensklinikum Linz GmbH Elisabethinen /ID# 247284, Linz, Upper Austria
  - Klinik Ottakring /ID# 247285, Vienna, Vienna
  - Hanusch Krankenhaus /ID# 247282, Vienna
- Switzerland (12):
  - Kantonsspital Aarau AG /ID# 251598, Aarau, Canton of Aargau
  - Kantonsspital Baden /ID# 241896, Baden, Canton of Aargau
  - Duplicate_Universitätsspital Basel /ID# 256509, Basel, Canton of Basel-City
  - Luzerner Kantonsspital /ID# 239242, Lucerne, Canton of Lucerne
  - Kantonsspital St. Gallen /ID# 239233, Sankt Gallen, Canton of St. Gallen
  - Hôpital du Chablais, Rennaz /ID# 241895, Rennaz, Canton of Vaud
  - KSW Kantonsspital Winterthur /ID# 239852, Winterthur, Canton of Zurich
  - Hirslanden Klinik /ID# 239239, Zurich, Canton of Zurich
  - EOC Ospedale Regionale di Bellinzona e Valli /ID# 240663, Bellinzona, Canton Ticino
  - Spitalzentrum Oberwallis /ID# 241897, Brig, Valais
  - Inselspital, Universitaetsspital Bern /ID# 239241, Bern
  - Hôpital de Nyon /ID# 240720, Nyon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info. — https://www.rxabbvie.com/